CLINICAL TRIAL: NCT02392975
Title: Fast MR for Young Children With Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-1917
Record Dates: First submitted 2015-03-02; First posted 2015-03-19 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: TBI (Traumatic Brain Injury)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fast magnetic resonance imaging (Fast MR) (Experimental): All subjects will undergo fast MR in addition to Computerized Tomography (CT) (the current criterion standard). Fast MR will be interpreted independently for research purposes by 2 blinded radiologists. Consensus interpretation will be compared to the clinical reading of the CT.
  Interventions: Procedure: Fast MR; Procedure: Computed Tomography

INTERVENTIONS:
Procedure: Fast MR — Enrolled subjects will undergo fast MR within 24 hours of CT completion. Subjects will be scanned using one of 2 Philips Ingenia MR 3T scanners. The estimated duration of the fast MR is less than 5 minutes, even if up to 2 sequences are repeated for motion.
  Other Names: Magnetic Resonance Imaging
Procedure: Computed Tomography — The Investigator will recruit children in whom a head CT is ordered as standard of care for TBI. Consenting subjects will undergo fast MR shortly after CT and results will be compared.

SUMMARY:
This proposal will test the diagnostic utility of fast magnetic resonance (MR) in young children with Traumatic brain Injury (TBI).

In children, TBI causes >2000 deaths, 35,000 hospitalizations and 470,000 emergency department visits in the US each year, making it a leading cause of pediatric disability and death. Currently 20-50% of these children undergo computed tomography (CT) scanning, exposing them to harmful radiation, and increasing their lifetime risk of cancer. Risks are especially increased in children because the neurologic exam is less reliable, because growing tissues are more vulnerable to radiation, and because children have more years to accumulate harmful mutations.

Fast MR is a short, motion-tolerant protocol that has been used in children with shunted hydrocephalus to eliminate radiation exposure without the need for sedation. However, fast MR has not been validated in children with TBI, a critical gap. The investigators will measure feasibility and diagnostic utility of fast MR in children < 6 years (72 months) old who undergo head CT for TBI.

The Investigator will recruit children in whom a head CT is ordered for TBI. Consenting subjects will undergo fast MR shortly after CT and results will be compared to determine: 1) whether fast MR identifies all traumatic injuries identified by CT and 2) whether fast MR without sedation can be performed quickly and successfully.

ELIGIBILITY:
Inclusion Criteria:

* Children <72 months old in whom a head CT is ordered/obtained with concerns for TBI
* Present to the Children's Hospital Colorado (CHCO) Emergency Department (ED) or inpatient wards

Exclusion Criteria:

* Contraindication to MR (e.g. pacemaker, implanted metallic object incompatible with MR)
* Prior diagnosis of TBI, structural brain lesion or prior brain surgery including shunted hydrocephalus
* Prior participation in this study
* Clinically unstable in the opinion of the patient's attending physician
* Wards of the State
* TBI not included in the differential diagnosis of the patient's attending physician (e.g. the indication for imaging is concern for infections, tumor, autoimmune or inflammatory disease) or if imaging has already identified a non-traumatic source for symptoms

Max Age: 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2015-06-02 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic utility (sensitivity/specificity) of fast MR to identify radiographic evidence of trauma as determined by dual, independent review by 2 masked pediatric neuroradiologists | 0-15 minutes
  The main outcome measure will be the identification of radiographically apparent brain injury using cranial CT as the gold standard. Diagnostic utility (sensitivity/specificity) of fast MR to identify radiographic evidence of trauma (yes/no) as determined by dual, independent review by 2 masked pediatric neuroradiologists and compared to the clinical interpretation of CT (the current criterion standard).

SECONDARY OUTCOMES:
Accuracy of fast MR to determine type and location of injury as determined by dual, independent review by 2 masked pediatric neuroradiologists and compared to the clinical interpretation of CT (the current criterion standard). | 0-15 minutes
Completion rate: determined by the number of fast MR's completed per protocol parameters (all sequences completed in <30 minutes; no request to stop imaging from physician, patient or family) | 0-5 minutes
Imaging time as determined by the time to complete all images - timer embedded in MR device | 0-5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: David M Lindberg, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado School of Medicine, Aurora, Colorado, United States

REFERENCES:
- [Derived] Lindberg DM, Stence NV, Grubenhoff JA, Lewis T, Mirsky DM, Miller AL, O'Neill BR, Grice K, Mourani PM, Runyan DK. Feasibility and Accuracy of Fast MRI Versus CT for Traumatic Brain Injury in Young Children. Pediatrics. 2019 Oct;144(4):e20190419. doi: 10.1542/peds.2019-0419. PMID 31533974